CLINICAL TRIAL: NCT04982536
Title: A Proof of Concept Assessment of the VMCore Biopsy System for Sampling and Retrieving Prostate Biopsy Cores Compared to a Standard of Care Biopsy
Brief Title: Assessment of VMCore Biopsy Versus Standard of Care Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uro-1 Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VMCore Assessment
Record Dates: First submitted 2021-07-15; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Each subject will have biopsy performed with both the study needle and a standard of care needle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- VMCore Biopsy System (Experimental): The VMCore biopsy needle will used to collect up to 10 tissue samples.
  Interventions: Device: VMCore Biopsy System
- Standard of Care Biopsy Needle (Active Comparator): The urologist will use his/her standard biopsy needle to collect up to 15 tissue samples.
  Interventions: Device: Standard of Care Biopsy Needle

INTERVENTIONS:
Device: VMCore Biopsy System — Prostate Examine
  Arms: VMCore Biopsy System
Device: Standard of Care Biopsy Needle — Prostate Examine
  Arms: Standard of Care Biopsy Needle

SUMMARY:
Prostate biopsy is the definitive test to establish the diagnosis of prostate cancer. The standard of care biopsy needles do not predictably obtain full cores of tissue and what tissue obtained is often fragmented, making pathologic review a challenge. The VMCore Biopsy System has a geometry in the tip of its biopsy needles that capture more tissue in a single sample. This study is to compare the characteristics of tissue captured by either standard of care needles and the VMCore needle.

DETAILED DESCRIPTION:
This post-market study is being conducted in order to assess the capability of the VMCore biopsy needle to capture prostate tissue in subjects consenting to the use of both the VMCore needle and the urological practice's standard of care needle for twinned samples during a routine prostate biopsy procedure. The primary endpoints are to success in tissue core sampling, safety of the sampling, and subject's tolerance to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Scheduled for a prostate biopsy
* Able and willing to provide verbal assessment of his condition 5 days post-procedure

Exclusion Criteria:

* Unable or unwilling to provide consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males have a prostate
Enrollment: 40 (Estimated)
Dates: Start 2020-07-19 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Procedure Success | 1 Day of the procedure
  Percentage of tissue samples suitable for pathological review
Adverse Events | 1 Day of the procedure
  Incidence and Severity of Adverse events associated with use of the biopsy needles
Patient Pain During use of the biopsy needles | 1 Day of the procedure
  Pain measured with Likert Scale of 1 to 5

SECONDARY OUTCOMES:
Mean Tissue volume for each sample taken | 1 Day of the procedure
  Length and diameter of tissue samples for cubic centimeters of volume

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lawson, Study Director — Uro-1 Medical
Locations (1):
- Georgia Urology, Cartersville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
No patient data will be shared among researchers. Tissue data may be shared